CLINICAL TRIAL: NCT06317285
Title: A Phase 2, Randomized, Double-Blind, Placebo Controlled, Parallel Group Study (TRANSFORM) to Evaluate the Efficacy and Safety of GSK3915393 in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Study to Evaluate the Efficacy and Safety of GSK3915393 in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study met futility criteria at pre-planned interim analysis, showing no clinical efficacy of the investigational drug. Based on the lack of efficacy at the interim data review, the sponsor decided to terminate the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 220929; 2023-509371-16-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: GSK3915393; Idiopathic Pulmonary Fibrosis; Efficacy; Safety; Forced vital capacity; Tolerability
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double-blind study with respect to allocation of GSK3915393 or placebo to participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK3915393 (Experimental): Participants will receive GSK3915393
  Interventions: Drug: GSK3915393
- Placebo (Experimental): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3915393 — GSK3915393 will be administered.
  Arms: GSK3915393
Drug: Placebo — Placebo will be administered.
  Arms: Placebo

SUMMARY:
Idiopathic Pulmonary Fibrosis is a chronic lung disease which causes scarring of the lungs and difficulty in breathing. GSK3915393 is a new medicine, which is being tested in participants with IPF for the first time. The study will assess the safety and effectiveness of GSK3915393 in IPF participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with IPF diagnosed within 5 years prior to screening based on the applicable American Thoracic Society (ATS)/ European Respiratory Society (ERS)/ Japanese Respiratory Society (JRS)/ Latin American Thoracic Society (ALAT) Guideline at the time of diagnosis.
* Centrally read chest High Resolution Computed Tomography (HRCT) obtained at screening or historical HRCT obtained within 12 months of screening that is consistent with Usual interstitial pneumonia (UIP) or probable UIP (if indeterminate HRCT finding, IPF may be confirmed locally by historical biopsy).
* FVC greater than or equal to (>=) 45 percent (%) of predicted normal.
* Diffusing Capacity (of Lung) for Carbon Monoxide (DLCO) >=25% of predicted normal corrected for hemoglobin (Hb).
* Prebronchodilator Forced Expiratory Volume in 1 second (FEV1)/FVC ≥ 0.7.
* If receiving antifibrotics must be on stable dose of nintedanib or pirfenidone for at least 12 weeks prior to screening.
* If not currently receiving pirfenidone or nintedanib, participant must have stopped pirfenidone or nintedanib for at least 4 weeks prior to screening.
* Body weight ≥40 kilogram (kg) and body mass index within the range 18.5-35 kilogram per meter square (kg/m2) (inclusive).
* A female participant is eligible to participate if a woman of nonchildbearing potential (WONCBP)
* Capable of giving signed informed consent

Exclusion Criteria:

* Participants with Interstitial Lung Disease (ILD) associated with other known causes.
* Diagnosis of sarcoidosis or any systemic autoimmune disease (including but not limited to scleroderma, polymyositis/dermatomyositis, systemic lupus erythematosus and rheumatoid arthritis).
* Acute IPF exacerbation within 6 months prior to screening and/or during the screening period (investigator-determined).
* Clinically significant non-parenchymal lung disease (e.g., asthma, chronic obstructive pulmonary disease, cavitary or pleural diseases) at screening.
* Diagnosis of severe pulmonary hypertension (investigator-determined)
* Extent of emphysema is greater than the extent of fibrosis according to reported results from the most recent HRCT.
* History of previous lung transplant or recent major surgery (investigator-determined) within 12 weeks prior to screening or planned during the trial period. Registration on a transplant waiting list is allowed.
* Clinically significant respiratory tract infection (e.g., active tuberculosis, infectious pneumonia, Corona virus disease 2019 [COVID-19]) requiring treatment within 4 weeks prior to and/or during the screening period.
* Cigarette smoking (including e-cigarettes) either current or within 3 months before screening.
* Current or chronic liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Alanine transaminase (ALT), Aspartate transaminase (AST), Alkaline phosphatase (ALP) >2x Upper Limit of Normal (ULN) and bilirubin >1.5x ULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than (<) 35% at screening).
* Clinically significant abnormalities detected on ECG of either rhythm or conduction, a Corrected QT interval (QTc) >450 millisecond (msec) or QTc > 480msec for participants with a bundle branch block and/or a pacemaker who are actively ventricularly pacing during the screening ECG.
* Participants with pacemakers who are not pacing at the time of the screening ECG should have a non-paced QTc <450 msec.

Prior/Concomitant Therapy-

* Simultaneous use of pirfenidone and nintedanib at screening.
* Received systemic corticosteroids equivalent to prednisone >10 mg/day or equivalent within 2 weeks of screening period.
* Use of any of the following therapies within 4 weeks prior to screening and during the screening period or planned during the study:
* Immunomodulatory therapies, including but not limited to azathioprine, mycophenolate mofetil, methotrexate, tacrolimus, cyclophosphamide, imatinib, Tumour Necrosis Factor -Alpha (TNF- α) inhibitors.
* Medications that are under investigation for the treatment of IPF including inhaled treprostinil and Phosphodiesterase-4 (PDE-4) inhibitors. Symptomatic cough therapies are allowed.
* Current use of systemic strong and moderate inducers or inhibitors of Cytochrome P450 3A4 (CYP3A4) (see prohibited medication section for further information) that cannot be safely discontinued or switched to an alternative agent at least 14 days before randomization.
* Current use of systemic CYP3A4 substrates that have a narrow therapeutic index that cannot be safely discontinued or switched to an alternative agent at least 14 days before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Absolute Change from Baseline in Forced Vital Capacity (FVC) in milliliters (mL) at Week 26 | Baseline and at Week 26

SECONDARY OUTCOMES:
Absolute Change from Baseline in Forced Vital Capacity (mL) at Weeks 4, 8, 12 and 18 | Baseline and at Week 4, Week 8, Week 12 and Week 18
Absolute Change from Baseline in Percent Predicted Forced Vital Capacity (%) at Weeks 4, 8, 12, 18 and 26 | Baseline and at Week 4, Week 8, Week 12, Week 18 and Week 26
Participants Achieving Relative Decline from Baseline in FVC (mL) Less than or Equal to (≤) 5 Percent (%) at Week 26 | Baseline and at Week 26
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 26
Number of Participants with Clinically Important Findings in Vital Signs | Baseline and Up to Week 26
Number of Participants with Clinically Important Findings in Electrocardiogram (ECG) | Baseline and up to Week 26
Number of Participants with Clinically Important Findings in Haematology | Baseline and up to Week 26
Number of Participants with Clinically Important Findings in Hepatobiliary Parameters | Baseline and up to Week 26
Number of Participants with Clinically Important Findings in Clinical Chemistry | Baseline and up to Week 26
Maximum observed concentration (Cmax) of GSK3915393 in IPF Participants | At Week 2 (pre-dose, and 0.5, 1, 1.5, 2, 3 and 4 hour (h) post-dose)
Area under the time-concentration curve (AUC) from Zero (pre-dose) to 4 hours (h) post-dose sample [0-4 h]) of GSK3915393 | At Week 2 (pre-dose, and 0.5, 1, 1.5, 2, 3 and 4 hour (h) post-dose)
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC- inf) of GSK3915393 | At Week 2 (pre-dose, and 0.5, 1, 1.5, 2, 3 and 4 hour (h) post-dose)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (54):
- United States (10):
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Cypress, Texas
- Argentina (6):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Florida
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Rosario
- Canada (5):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Trois-Rivières, Quebec
- France (6):
  - GSK Investigational Site, La Tronche
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Toulouse
- Germany (4):
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Heidelberg
  - GSK Investigational Site, Wuppertal
- Italy (9):
  - GSK Investigational Site, Catania
  - GSK Investigational Site, Monza MB
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Perugia
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Sassari
  - GSK Investigational Site, Torrette AN
- Netherlands (2):
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Rotterdam
- Poland (3):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Poznan
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
- United Kingdom (3):
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Leeds West Yorkshire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/